CLINICAL TRIAL: NCT03594084
Title: Retrospective Clinical Study of Malaria in Strasbourg University
Brief Title: Malaria in Strasbourg University Hospital
Acronym: ACMUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7084
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-07

CONDITIONS: Malaria
Keywords: Malaria; Malaria imported cases; Recurrent malaria; Endemic malaria areas; Biological diagnosis; Hospital vs private laboratory diagnosis
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary purpose is to describe the anamnestic, clinical, biological, and therapeutic characteristics of imported malaria in people originated from endemic areas. Indeed, clinicians have observed that people from such areas start malaria just after their arrival in France. Such observation needed to be confirmed. In addition, The investigators observed a variation in the laboratory diagnostic performance of malaria between hospital and private laboratories. Such observation also needed to be analyzed objectively

ELIGIBILITY:
Inclusion Criteria:- Patient over 18 years

* Patients from birth to 18 years
* Patient submitted to guardianship
* Patient submitted to trusteeship
* Diagnosis patients with malaria from 01/01/2017 to 01/01/2018
* Patient or legal representative agree to use medical data for this research

Exclusion Criteria:

* Lack of confirmation malaria diagnosis
* Impossibility to inform patients
* Patient who does not wish to participate in the study
* Patient submitted to justice safeguarding

Min Age: 1 Day | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: iagnosis patients with malaria from 01/01/2017 to 01/01/2018
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Study of clinical characteristics of imported malaria in people originated from endemic areas hospitalized at Strasbourg University Hospital from 2017 to 2018. | The period from January 1st, 2017 to January 1st, 2018 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Xavier ARGEMI, MD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Maladies Infectieuses et Tropicales, Strasbourg, France